CLINICAL TRIAL: NCT04323475
Title: A Randomized, Open-Label, Active Controlled Study to Evaluate the Safety and Tolerability of a Phage Cocktail-SPK Therapy in Second Degree Burn Wounds in Adult Patients
Brief Title: Phage Therapy for the Prevention and Treatment of Wound Infections in Burned Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Precisio Biotix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGX-18001
Record Dates: First submitted 2020-03-20; First posted 2020-03-26 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Wound Infection
Keywords: Burns; Infection; Infection wound; Infection, Bacterial; Infection Pseudomonas Aeruginosa; Infection Staphylococcus Aureus; Infection, Klebsiella pneumoniae; Resistant Infection
MeSH Terms: conditions — Wound Infection; Burns; Infections; Bacterial Infections; Pseudomonas Infections; Staphylococcal Infections | interventions — 2,4,6-tribromophenol; Gramicidin, Neomycin Sulfate, Nystatin, Triamcinolone Acetonide Drug Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care consists of Xeroform primary dressing, a Melolin interface and a crepe. Kenacomb will be used for participants with diagnosed or suspected local infections.
  Interventions: Drug: Xeroform
- Cocktail-SPK and standard of care (Experimental): The experimental drug consists of Cocktail-SPK used as an adjunct to the standard of care. Standard of care consists of Xeroform primary dressing, a Melolin interface and a crepe. Kenacomb will be used for participants with diagnosed or suspected local infections.
  Interventions: Biological: Bacteriophage cocktail spray; Drug: Xeroform

INTERVENTIONS:
Biological: Bacteriophage cocktail spray — Study intervention consists of a dosage-metered airless spray containing a cocktail of 14 bacteriophages at a concentration of 1.4 x 10^8 PFU/mL for an effective dosage of 2.5 x10^5 PFU/cm^2 of burned area. The study intervention will be applied in conjunction with standard of care.
  Other Names: PGX-0100; Phage cocktail-SPK
  Arms: Cocktail-SPK and standard of care
Drug: Xeroform — Standard of care will consist of Xeroform primary dressing and Kenacomb topical antibiotic cream (for wounds with signs of localized infection)
  Other Names: Kenacomb

SUMMARY:
The central aim of this trial is to investigate the safety and tolerability of Phage Cocktail-SPK as an adjunct to standard therapy for the prevention and treatment of burns susceptible to infection/or infected by S. aureus, P. aeruginosa, or K. pneumoniae species. It is hypothesized that no adverse events, clinical abnormalities, or changes in laboratory tests results related to the application of Phage Cocktail SPK Spray will be observed.

DETAILED DESCRIPTION:
This is a Phase I, randomized, open-label, active controlled study to evaluate the safety and tolerability of a Phage Cocktail-SPK therapy for second degree burn wounds in adult patients. The wound will be clinically selected on the basis that it is a second degree burn less than 10 percent of total body surface area, and that, according to medical assessment, should heal without surgical intervention. The study is intended to include one site outside of the United States of America, namely the Royal Brisbane and Women's Hospital, in Brisbane, Queensland, Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and lifestyle considerations, and availability for the duration of the study
3. Male or female, aged 18 years or older presenting at the emergency department, out-patient burn department or in-hospital patients with a thermal second degree burn wounds (American Burn Association severity classification).
4. Patients with a burn wound covering less than 10% of their total body surface area (TBSA) and present within 7 days of their injury, with or without signs of local infection, expected to heal without the need for surgery.
5. For females of reproductive potential: use of a highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of administration of the study intervention
6. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

1. Current use of dressings containing silver or nanocrystalline silver
2. Pregnancy or lactation
3. Clinical evidence of invasive infection based on American Burn Association consensus conference(Greenhalgh et al., 2007).
4. Burn wounds present in anatomic locations such as burns on the face, hands, feet, genitals, perineum, as well as sites at high risk for developing compartment syndrome (deep circumferential extremity burns).
5. Known allergic reactions to components of Xeroform or Kenacomb.
6. Patients diagnosed with Type I or Type II diabetes.
7. Treatment with another investigational drug or other intervention within 30 days
8. Intercurrent condition requiring a high dose of chronic corticosteroid therapy, immunosuppressive medication, oncologic chemotherapy.
9. Patients who have additional uncontrolled serious medical or psychiatric illness determined by the investigators where the patient is unfit to receive PGX-0100.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events coded by MedDra | At least 14 days
  Safety of Phage cocktail-SPK will be measured by the number and percent of treatment related adverse events
Incidence of treatment discontinuation due to adverse events | 14 days
  Tolerability of Phage Cocktail-SPK will be measured by the percent premature discontinuation from the study intervention due to treatment emergent Adverse Events

SECONDARY OUTCOMES:
Assess if Phage Cocktail-SPK can prevent or reduce S. aureus, P. aeruginosa, or K. pneumoniae wound colonization. | 14 days
  Change in the incidence of positive wound cultures for S. aureus, P. aeruginosa, K. pneumoniae;

OTHER OUTCOMES:
Determine the effect of Phage Cocktail-SPK treatment on burn wound progression. | 14 days
  Rate of wound re-epithelization by visual judgment and burn depth and progression by photography.
Determine the effect of Phage Cocktail-SPK treatment on the sensitivity profiles of S. aureus, P. aeruginosa, or K. pneumoniae present in the wound | 14 days
  Change in antibiotic and phage sensitivity profile of S. aureus, P. aeruginosa, K. pneumoniae.
Assess the production of phage antibodies | 14 days
  Presence of Phage Cocktail-SPK antibodies in serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Tawil, PhD, Study Director — Precisio Biotix Therapeutics, Inc.